CLINICAL TRIAL: NCT01466972
Title: Reversing Hormone Resistance in Advanced Breast Cancer With Pazopanib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hope Rugo, MD (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Hope Rugo, MD, Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 117513; NCI-2012-00494 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2011-10-25; First posted 2011-11-08 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer; Breast Neoplasm
Keywords: Advanced; Breast; Cancer; Hormone Resistance; Pazopanib; anastrozole; arimidex; letrozole; femara
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pazopanib in combination with a NSAI (Experimental): Non-randomized, open label
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Oral, 800mg tablet daily per cycle
  Other Names: Votrient

SUMMARY:
The purpose of this study is to evaluate the clinical benefit rate at 12 weeks from the addition of pazopanib to a non-steroidal aromatase inhibitor (NSAI) (letrozole or anastrozole) in patients with hormone receptor positive advanced breast cancer progressing on the same NSAI hormone therapy.

DETAILED DESCRIPTION:
In this trial, the investigators propose to evaluate the role of VEGFR blockade with the tyrosine kinase inhibitor pazopanib in combination with nonsteroidal aromatase inhibitors (NSAI) in patients who are progressing or have relapsed on the same NSAI hormone therapy given for advanced or early stage breast cancer. If this trial demonstrates clinical benefit, this all oral combination could be tested in both the neoadjuvant and metastatic settings in a randomized phase II design.

In order to investigate potential factors predicting response or resistance to pazopanib and NSAIs, several translational studies have been incorporated into this trial.

The prognostic value of circulating tumor cells (CTC) has been demonstrated in several studies in breast cancer, especially in advanced stage [35-38]. At University of California, San Francisco (UCSF) in the laboratory of Dr. John Park, the investigators have demonstrated expertise in the measurement of CTC in patients with advanced stage breast cancer by IC/FC assay. CTC are first enriched with immunomagnetic beads coated with EpCAM, then EpCAM+, CD45-, nucleic acid+ cells are detected by flow cytometry. This technique is highly sensitive and reproducable, and allows sorting of cells for molecular analysis as well as analysis of cell surface markers[39]. In this trial, the investigators will collect patient's peripheral blood samples every 4 weeks while on treatment and follow any reduction of CTC.

The mechanisms of hormonal resistance includes intrinsic and acquired pathways: decreased ER expression accounts for intrinsic resistance and the increased receptor tyrosine kinase pathway relates to acquired resistance [40-42]. The investigators plan to analyze the mutation of PI3K/Akt and deletion of PTEN by sequencing in CTC (depending on numbers of cells, which in turn determines feasibility), in order to make a preliminary assessment of potential markers of response to pazopanib.

The tumor microenvironment plays an important role in cancer development and progression. Clinical studies have revealed that the increased T regulatory cells (Treg), high ratios of CD4/CD8 T lymphocytes, and extra follicular B cells in primary tumors correlated with worse overall survival [43-45]. Recently, studies from preclinical models have shown that tumor associated macrophages (TAM) can promote pulmonary metastases in breast cancer animal models, and in both the preclinical and clinical settings are associated with worse clinical outcome [46-48]. TGFβ has been linked to hormonal resistance in breast cancer. The activation of TGFβ leads to increased regulatory CD4+ T cells and decreased cytotoxic CD8+ T cells in the tumor microenvironment [49]. A recent study in non-small cell lung cancer suggests that baseline and post-treatment levels of cytokines, particularly IL-4 and IL-12 correlated with response to pazopanib[50]. In this study, the investigators will collect patient's serum to monitor the level of cytokines at baseline and during treatment, the investigators will compare the change of cytokine level with pazopanib in each patient, and also compare between responders and non-responders. This information may help us to identify biomarkers that would predict response to antiangiogenic therapy and to identify possible mechanisms of resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to performance of study specific procedures or assessments, and must be willing to comply with treatment and follow up.

   - Procedures conducted as a part of routine clinical management of the subject (e.g., blood count, imaging study) and obtained prior to signed informed consent may be utilized for Screening or Baseline purposes provided these tests are obtained as specified in the protocol).
2. Subjects must have measurable or evaluable disease. Disease sites that are evaluable for progression but not measurable per RECIST guidelines include:

   * Bone lesions
   * Previously irradiated lesions
   * Cutaneous manifestations (non-discreet lesions only)
3. Age ≥ 18 years.
4. Postmenopausal women defined by one of the criteria:

   * No spontaneous menses for at least 12 months if the subject is ≥ 50 years old;
   * Amenorrheic for at least 12 months if the subject is < 50 years old, with serum estradiol within the institutional postmenopausal range;
   * Bilateral oophorectomy;
   * If prior hysterectomy but intact ovaries, must be ≥ 55 years old, or have serum estradiol within the postmenopausal range;
   * If premenopausal, must be on a GnRH agonist (leuprolide or goserelin) with serum estradiol levels within the institutional postmenopausal range.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2.
6. Histologically or cytologically confirmed estrogen receptor (ER) and/or progesterone receptor (PgR) positive carcinoma of the breast with unresectable, locally advanced and/or metastatic (AJCC Stage IV) disease.
7. Subjects must have received prior hormonal therapy for the treatment of breast cancer as follows:

   * Progression must be documented while taking a nonsteroidal aromatase inhibitor including anastrozole or letrozole.
   * No more than 2 prior hormonal therapies for metastatic disease.
   * If hormonal therapy was administered in the adjuvant setting, subjects must have received therapy for at least 6 months prior to developing metastatic disease.

   Note: A regimen of sequential tamoxifen/AI in the adjuvant setting is considered to be one therapy

   - If hormonal therapy was administered in the metastatic setting, subjects must have received therapy for at least 3 months prior to progression
8. Subjects whose tumors overexpress ErbB2 are eligible provided that they have progressed following therapy which included trastuzumab and/or lapatinib.

   Note for prior lapatinib: Subjects must have completed therapy with lapatinib at least 7 days prior to the first dose of study drug.

   Note for prior trastuzumab: Subjects who received Q3 weekly, Q2 weekly or Q1 weekly must have completed therapy with trastuzumab at least 3 weeks, 2 weeks or 1 week, respectively, prior to the first dose of study drug.
9. Adequate hematologic and hepatic function as defined in Protocol Table 1
10. Subjects must have discontinued hormone replacement therapy (HRT) (e.g., conjugated estrogens tablets, USP or premarin), at least 28 days prior to receiving the first dose of randomized therapy.
11. Radiotherapy prior to initiation of therapy is allowed to a limited area (e.g., palliative treatment for painful bone metastases), if it is not the sole site of disease. Subjects must have completed treatment at least one week prior to starting study drugs, and must have recovered from all treatment-related toxicities.
12. Bisphosphonate or RANK ligand inhibitor therapy for bone metastases is allowed. Prophylactic use of bisphosphonates in subjects without bone disease, except for the treatment of osteoporosis, is not permitted;
13. Ability to swallow and retain oral medication.

Exclusion Criteria:

1. Prior use of pazopanib
2. Premenopausal levels of estradiol, or ongoing menses (see definitions of menopause above).
3. Known central nervous system (CNS) metastases or leptomeningeal carcinomatosis. Screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if the subject has clinical findings suggestive of CNS metastasis.
4. History of another active malignancy. Note: Subjects who have had another malignancy and have been disease-free for 5 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
5. Clinically significant gastrointestinal abnormalities which might interfere with oral dosing, including, but not limited to:

   * Malabsorption syndrome
   * Major resection of the stomach or small bowel that could affect the absorption of study drug
   * Inflammatory bowel disease
   * Ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation
   * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment
6. Presence of uncontrolled infection.
7. Prolongation of corrected QT interval (QTc) >480msecs.
8. History of any one or more of the following cardiovascular conditions within the past 6 months:

   * Angioplasty or stenting
   * Myocardial infarction
   * Unstable angina
   * Coronary artery by-pass graft surgery
   * Symptomatic peripheral vascular disease
9. Class II, III or IV congestive heart failure, as defined by the New York Heart Association (NYHA).
10. Use of an investigational agent, including an investigational anti-cancer agent, within 14 days prior to the first dose of study drug.
11. Prior use of an investigational drug that targets VEGF or VEGF receptors.
12. Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 and/or that is progressing in severity.
13. Poorly controlled hypertension (defined as systolic blood pressure (SBP) of ≥140mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg).

    Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. Blood pressure must be re-assessed prior to start of study therapy. The mean SBP/DBP values must be <140/90mmHg (OR 150/90mmHg, if this criterion is approved by Safety Review Team) in order for a subject to be eligible for the study.
14. History of cerebrovascular accident (CVA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.

    Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulant agents for at least 6 weeks are eligible.
15. Major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer not related to cancer (procedures such as catheter placement not considered to be major).
16. Evidence of active bleeding or bleeding diathesis.
17. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04-27 (Actual); Primary Completion 2015-12-07 (Actual); Study Completion 2019-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hope Rugo, M.D., Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pazopanib in Combination With a NSAI
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pazopanib in Combination With a NSAI
Number analyzed (Participants) | 30
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 4
  50-59 years | 13
  60-69 years | 9
  70-79 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Benefit (CB)
Description: For the purpose of this study, participants who obtained a complete response (CR), partial response (PR), or stable disease (SD) at 12 weeks per Response Evaluation Criteria in Solid Tumors (RECIST) guidelines version 1.1 were defined as having a clinical benefit from the treatment. An overall response rate of 20% was considered to be clinically meaningful. All participants who take at least two weeks of study drug and the non-steroidal aromatase inhibitor were evaluated for toxicity and efficacy
Time Frame: 12 weeks
Population: Twenty-eight patients met the 2 weeks of treatment minimum needed to be considered evaluable for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib in Combination With a NSAI
Number analyzed (Participants) | 28
Participants | 13

2. Secondary Outcome: Progression Free Survival
Description: Evaluate progression free survival with ongoing evaluations at 12 week intervals until progression or up to 2 years, whichever is first.
Time Frame: up to 2 years
Population: Twenty-eight patients met the 2 weeks of treatment minimum needed to be considered evaluable for this endpoint.
Measure: Median (Full Range); unit: weeks
Arm/Group | Pazopanib in Combination With a NSAI
Number analyzed (Participants) | 28
weeks | 20 [2 to 104]

3. Secondary Outcome: Number of Participants Experiencing Any Treatment-related Adverse Events (AE)
Description: All patients who take at least two weeks of study drug and the non-steroidal aromatase inhibitor will be evaluable for treatment-related toxicity by ongoing evaluations at 4 week intervals until progression or up to 2 years, whichever is first.
Time Frame: up to 2 years
Population: Twenty-eight patients met the 2 weeks of treatment minimum needed to be considered evaluable for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib in Combination With a NSAI
Number analyzed (Participants) | 28
Participants | 26

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Pazopanib in Combination With a NSAI
All-Cause Mortality (participants affected / at risk) | 2/30
Serious Adverse Events (participants affected / at risk) | 8/30
Other Adverse Events (participants affected / at risk) | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pazopanib in Combination With a NSAI (N=30)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pazopanib in Combination With a NSAI (N=30)
Nausea (Gastrointestinal disorders) | 15 (21)
Diarrhea (Gastrointestinal disorders) | 11 (13)
Abdominal pain (Gastrointestinal disorders) | 7 (11)
Vomiting (Gastrointestinal disorders) | 5 (10)
Constipation (Gastrointestinal disorders) | 4 (7)
Dry Mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (3)
Fatigue (General disorders) | 16 (21)
Chills (General disorders) | 3 (4)
Fever (General disorders) | 2 (3)
Non-cardiac chest pain (General disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Hypertension (Vascular disorders) | 9 (11)
Hot flashes (Vascular disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 9 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (9)
Headache (Nervous system disorders) | 5 (7)
Dysgeusia (Nervous system disorders) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 5 (9)
Alanine aminotransferase increased (Investigations) | 4 (11)
Investigations - Other (Investigations) | 4 (24)
Alkaline phosphatase increased (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (9)
Platelet count decreased (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 2 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Blurred vision (Eye disorders) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 2 (3)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (5)
Hypothyroidism (Endocrine disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT01466972/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2017-07-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT01466972/Prot_SAP_002.pdf